CLINICAL TRIAL: NCT01501422
Title: Effect of Estrogen Therapy on Objective Sleep Quality in Postmenopausal Women at Menopause Clinic, King Chulalongkorn Memorial Hospital, Double- Blind, Randomized, Placebo-controlled Trial
Brief Title: Effect of Estrogen Therapy on Objective Sleep Quality in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pimpika Tansupswatdikul, MD., Principle investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRU CU-1/2011
Record Dates: First submitted 2011-11-14; First posted 2011-12-29 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Insomniac Postmenopausal Women
Keywords: postmenopause; sleep quality; estrogen; objective sleep quality; actigraph
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estrogen (Experimental): Use estrogen patch for 8 weeks
  Interventions: Drug: Estrogen patch
- Placebo (Experimental): Use placebo patch for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estrogen patch — 50 microgram estrogen patch weekly
  Arms: Estrogen
Drug: Placebo — Placebo patch for 8 weeks
  Arms: Placebo

SUMMARY:
1. Sex hormone including estrogen have synergistic effect to serotonin activity and decrease activity of monoamine oxidase activity so the norepinephrine is not be metabolized, these substance are important to regulate hemostasis and circadian process of sleep
2. Estrogen also regulate gamma-aminobutyric acid (GABA) secretion

   * GABA substance is in order to initiate sleep and continue sleep
3. According to epidemiologic data, problem of sleep was increasing in postmenopause group compare to premenopause group (aged-match)
4. This research perform to find out the actual effect of estrogen in improving sleep quality.

DETAILED DESCRIPTION:
1. 40-60 year-old postmenopausal women with insomnia and mild-moderate vasomotor symptom were screened and included in project
2. Block of four randomization was use to categorize participants into 2 groups

   * Study group (estrogen patch)
   * Control group (placebo patch)
3. Sleep quality was measured before intervention by subjective and objective sleep quality

   * Subjective sleep quality (self sleep questionnaire)
   * Objective sleep quality (wrist actigraphy and sleep diary):

   wrist actigraph sleep test at home for 1 week
4. Intervention phase : continuous use of weekly patch for 8 weeks

   * Estrogen patch in study group
   * Placebo patch in control group
5. Follow up phase

   * At 4 weeks of use, investigator will telephone call for follow up the participant's compliance and the side effects during patch use.
   * After completed use of 7th patch, sleep quality was measured again, self sleep quality questionnaire and 1 week-wrist actigraphy and sleep diary test
6. Then the data will be analysed and open label, in nonhysterectomized postmenopausal women in study group will take the medroxyprogesterone acetate for washing out the endometrium for 2 weeks
7. The participants will be counseled, further investigate and proper treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women 40-60 years old
* Mild to moderate vasomotor symptom
* Insomnia
* fluent read and write in Thai language
* Inform consent

Exclusion Criteria:

* Acute liver and gall bladder disease
* undiagnosed abnormal bleeding per vagina
* History of BIRADs 3 from mammogram
* History or current venous thrombosis, embolism
* diagnosis of sleep disorder
* use of hypnotic drug or antihistamine in the past month
* Diagnosis of psychiatric disorder such as depressive disorder, schizophrenia, anxiety disorder
* No past history of malignancy
* No history of chronic renal disease, alzheimer's disease, uncontrolled hypertension, uncontrolled diabetes mellitus
* history of estrogen use in past 6 months
* drug abuse, Alcohol

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (SE) | 8 months
  Sleep efficiency is proportion of sleep in the period potentially filled by sleep-ratio of total sleep time to time in bed.

SECONDARY OUTCOMES:
Sleep latency (SL) | 8 months
  Sleep latency is the time period measured from "lights out," or bedtime, to the beginning of sleep.
Total sleep time (TST) | 8 months
  TST is amount of actual sleep time in a sleep period.
Wake time after sleep onset (WASO) | 8 months
  WASO is the total time of awake occurring between sleep onset and final wake up.
Number of awakening | 8 months
  Number of awakening is the number of awakening during onset of sleep and final wake-up.
Score of two sleep quality assessment questionnaires. | 8 months
  * Insomnia severity index is the 7 topic questionnaire for determine the severity of insomnia problem.
  * Ebworth severity index is the questionnaire to assess daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Pimpika Tansupswatdikul, MD., Principal Investigator — Chulalongkorn University; Sukanya Chaikiitisilpa, MD., Study Chair — Chulalongkorn University
Locations (1):
- Menopause Clinic, Menopause research unit, King Chulalongkorn Memorial Hospital, Pathumwan, Bangkok, Thailand

REFERENCES:
- [Background] Kalleinen N, Polo O, Himanen SL, Joutsen A, Polo-Kantola P. The effect of estrogen plus progestin treatment on sleep: a randomized, placebo-controlled, double-blind trial in premenopausal and late postmenopausal women. Climacteric. 2008 Jun;11(3):233-43. doi: 10.1080/13697130802112033. PMID 18568788
- [Background] Huang KE, Baber R; Asia Pacific Tibolone Consensus Group. Updated clinical recommendations for the use of tibolone in Asian women. Climacteric. 2010 Aug;13(4):317-27. doi: 10.3109/13697131003681458. PMID 20443720
- [Background] Halbreich U, Kahn LS. Role of estrogen in the aetiology and treatment of mood disorders. CNS Drugs. 2001;15(10):797-817. doi: 10.2165/00023210-200115100-00005. PMID 11602005
- [Background] Shanafelt TD, Barton DL, Adjei AA, Loprinzi CL. Pathophysiology and treatment of hot flashes. Mayo Clin Proc. 2002 Nov;77(11):1207-18. doi: 10.4065/77.11.1207. PMID 12440557
- [Background] Sarti CD, Chiantera A, Graziottin A, Ognisanti F, Sidoli C, Mincigrucci M, Parazzini F; Gruppo di Studio IperAOGOI. Hormone therapy and sleep quality in women around menopause. Menopause. 2005 Sep-Oct;12(5):545-51. doi: 10.1097/01.gme.0000172270.70690.5e. Epub 2005 Sep 1. PMID 16145308
- [Background] Wiklund I, Berg G, Hammar M, Karlberg J, Lindgren R, Sandin K. Long-term effect of transdermal hormonal therapy on aspects of quality of life in postmenopausal women. Maturitas. 1992 Mar;14(3):225-36. doi: 10.1016/0378-5122(92)90117-m. PMID 1508062
- [Background] Polo-Kantola P, Erkkola R, Helenius H, Irjala K, Polo O. When does estrogen replacement therapy improve sleep quality? Am J Obstet Gynecol. 1998 May;178(5):1002-9. doi: 10.1016/s0002-9378(98)70539-3. PMID 9609575
- [Background] Saletu B. Sleep, vigilance and cognition in postmenopausal women: placebo-controlled studies with 2 mg estradiol valerate, with and without 3 mg dienogest. Climacteric. 2003 Aug;6 Suppl 2:37-45. PMID 14669843
- [Background] Ensrud KE, Stone KL, Blackwell TL, Sawaya GF, Tagliaferri M, Diem SJ, Grady D. Frequency and severity of hot flashes and sleep disturbance in postmenopausal women with hot flashes. Menopause. 2009 Mar-Apr;16(2):286-92. doi: 10.1097/gme.0b013e31818c0485. PMID 19002015
- [Background] Tranah GJ, Parimi N, Blackwell T, Ancoli-Israel S, Ensrud KE, Cauley JA, Redline S, Lane N, Paudel ML, Hillier TA, Yaffe K, Cummings SR, Stone KL. Postmenopausal hormones and sleep quality in the elderly: a population based study. BMC Womens Health. 2010 May 4;10:15. doi: 10.1186/1472-6874-10-15. PMID 20441593
- [Derived] Tansupswatdikul P, Chaikittisilpa S, Jaimchariyatam N, Panyakhamlerd K, Jaisamrarn U, Taechakraichana N. Effects of estrogen therapy on postmenopausal sleep quality regardless of vasomotor symptoms: a randomized trial. Climacteric. 2015 Apr;18(2):198-204. doi: 10.3109/13697137.2014.964670. Epub 2014 Nov 27. PMID 25242569